CLINICAL TRIAL: NCT03458936
Title: Resilience in Adolescent Development
Acronym: RAD
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor of Psychiatry, University of Texas Southwestern Medical Center
Other Study IDs: STU 062016-042
Record Dates: First submitted 2017-04-05; First posted 2018-03-08 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Risk Assessment; Resilience, Psychological; Depression; Mood Disorders; Anxiety Disorders; Mental Health
Keywords: Depression; Adolescence; Resilience; Risk Factor; Biomarker
MeSH Terms: conditions — Depression; Mood Disorders; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Urine, Saliva, Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individual at risk for a Mood Disorder: Youth aged 10-24, male and female of all races and ethnicity with either: a) a personal history (anxiety disorder, conduct disorder, substance use disorder, etc.) of a mental health disorder that is a not a mood disorder, OR b) no current or past mood disorder, but with Biological Family history (ex. mother, father, siblings, uncles, aunts, etc.) of mood disorder, substance use disorder, suicide deaths or attempts, or other mental health disorder.
- Healthy Individual: Youth aged 10-24, male and female of all races and ethnicity with no psychiatric diagnoses (no history of mood disorders and having no relative with a history of a mood disorder).

SUMMARY:
RAD is a 10-year natural history, longitudinal, prospective assessment study of a cohort of 2,500 participants (ages 10-24 years) that will help uncover the socio-demographic, lifestyle, clinical, psychological, and neurobiological factors that contribute to resilience among children, adolescents, and young adults at-risk for mood and anxiety disorders. As this is an exploratory study, we will assess a comprehensive panel of carefully selected participant specific parameters, including socio-demographic, life habits, clinical, biological, behavioral, neurophysiological, and neuroimaging. The study is designed to observe and collect factors associated with resilience in a non-invasive fashion; no interventions or treatments will be conducted during the project. Assessments will be conducted up to 4 times per year for up to 10 years, as well as a baseline visit. Study visits will be conducted in person whenever feasible but may be completed by phone/mail/computer, if an in-person visit is not possible.

DETAILED DESCRIPTION:
The primary objective of this initiative is identify and validate biosignatures of resilience. Specifically, the research will identify protective factors (socio-demographic, lifestyle, clinical and behavioral assessments, fluid-based biomarkers, genomics, neuroimaging, EEG, and cell-based assays) that reduce risk of developing mood and anxiety disorders in adolescents and young adults at risk for these illnesses.

Presence and severity of symptoms will be assessed over 10 years using questionnaires for symptom changes, social factors, and overall quality of life. Other outcomes generated from this study will include rate of change in quantitative measures of brain function, of depression relevant brain regions correlated with systems-levels behavior and other functional neuro-circuitry MRI measures. Rate of change of specified biochemical biomarkers will also be assessed. Integration of these measures will provide an unmatched understanding into the mechanisms of resilience and protection against depression and anxiety disorders and holds tremendous promise for identifying targets for prevention strategies.

Specific Aims of the RAD Study:

Aim 1 - Examine baseline biosignatures and independent factors (demographic, social, environmental, genetic, EEG, and fMRI) associated with resilience in at-risk adolescents and young adults.

Aim 2 - Examine changes in the biomarker factors annually for 10 years to determine for plasticity of these biomarkers.

Aim 3 - Examine the interaction between psychiatric symptoms and changes in the biopsychosocial signature.

Aim 4 - Evaluate psychological, social, and physiological correlates, from mobile based data, of mood changes to construct a model of risk and resilience to depression and mood disorders among adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

1. Youth aged 10-24, male and female of all races and ethnicity.
2. Able to speak, read, and understand English. However, the parent(s)/guardian(s)/legally authorized representatives (LAR) may either speak English or Spanish as the consenting process can be conducted bilingually.
3. Adults aged 18 and older must be able to provide written informed consent; for youth younger than age 18, parent(s)/guardian(s)/LAR must provide written informed consent, and the youth must provide written informed assent.
4. Ability to complete clinical evaluations and neuropsychological testing.
5. Belong to one of the following groups:

   1. Individual at risk for a Mood Disorder: defined as either: a) Personal history (anxiety disorder, conduct disorder, substance use disorder, etc.) of a mental health disorder that is a not a mood disorder, OR b) No current or past mood disorder, but individual with Biological Family history (ex. mother, father, siblings, uncles, aunts, etc.) of mood disorder, substance use disorder, suicide deaths or attempts, or other mental health disorder.
   2. Healthy Individual: defined as having no psychiatric diagnoses (no history of mood disorders and having no relative with a history of a mood disorder).

Exclusion Criteria:

1. Individuals who are unable to provide informed consent or assent.
2. Participants who are non-English speaking.
3. Individuals with any of the following psychotic features: Mood Disorder with psychotic features, schizophrenia, schizoaffective disorder, or other psychotic disorder.
4. (participants who develop depression during the longitudinal follow-up will continue in the study).
5. A PHQ-9 score of 10 or greater.
6. Individuals who are unable to provide a stable home address and contact information.
7. Has any condition for which, in the opinion of the investigator or designee, study participation would not be in their best interest (including but not limited to cognitive impairment, unstable general medical condition, intoxication, active psychosis) or that could prevent, limit, or confound the protocol-specified assessments.

Exclusion for Healthy Controls

1. A lifetime or a current history of a mood disorder based upon a semi-structured diagnostic interview.
2. Personal (anxiety disorder, conduct disorder, substance use disorder, etc.) history of a mental health disorder that is not a mood disorder, or Biological Family (ex. mother, father, siblings, uncles, aunts, etc.) with history of mood disorder, substance use disorder, suicide deaths or attempts or other mental health disorder. (May participate in the RAD study as a non-healthy control).
3. Meets any exclusion criteria as part of the main RAD study.

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be males or females between ages 10 and 24 who have provided informed consent.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-08-17 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Depression Severity | 10 Years
  Longitudinal changes in depression presence and severity of participants without a mood disorder on Patient Health Questionnaire (PHQ-9).
  Interpretation of Total Scores:
  0-4: Minimal depression or no depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-27: Severe depression

SECONDARY OUTCOMES:
Functioning (MRI) | 10 Years
  Comparison of Longitudinal changes in functioning as measured by Magnetic Resonance Imaging (MRI) in participants without a mood disorder.
Functioning (EEG) | 10 Years
  Comparison of Longitudinal changes in functioning as measured by quantitative electroencephalography (EEG) in participants without a mood disorder.
Biomarkers (Proteomic Methods) | 10 Years
  Comparison of longitudinal changes in fluid-based biomarkers as measured by proteomic methods in participants without a mood disorder.
Biomarkers (Metabolomics Methods) | 10 Years
  Comparison of longitudinal changes in fluid-based biomarkers as measured by metabolomics methods in participants without a mood disorder.
Biomarkers (Transcriptomic Methods) | 10 Years
  Comparison of longitudinal changes in fluid-based biomarkers as measured by transcriptomic methods in participants without a mood disorder.
Biomarkers (Genomic Methods) | 10 Years
  Comparison of longitudinal changes in fluid-based biomarkers as measured by genomic methods in participants without a mood disorder.
Biomarkers (Epigenomic Methods) | 10 Years
  Comparison of longitudinal changes in fluid-based biomarkers as measured by epigenomic methods in participants without a mood disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H. Trivedi, MD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided